CLINICAL TRIAL: NCT00105053
Title: A Phase I/II Study of an Antitumor Vaccination Using Alpha (1,3) Galactosyltransferase Expressing Allogeneic Tumor Cells in Patients With Hormone Refractory Prostate Cancer
Brief Title: Vaccine Treatment for Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Nicholas N. Vahanian, M.D., Chief Medical and Operations Officer, NewLink Genetics Corporation
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG0103; 398-04FB
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vaccine group (Experimental)
  Interventions: Biological: HyperAcute-Prostate Cancer Vaccine

INTERVENTIONS:
Biological: HyperAcute-Prostate Cancer Vaccine — Before enrollment in the Phase I and Phase II- Arm A studies, the patient must be determined to have measurable disease with biopsies on first recurrence or bone metastases. In the Phase II- Arm B study, patients will be men with non-measurable progressive disease as evidenced by elevated PSA only. Cells will be injected intradermally every two weeks for 12 cycles on a prime-boost regimen. Dosage will vary from 30 million to 500 million HAP cells.

SUMMARY:
This 2-phase study will determine the safety of treating patients with prostate cancer with the genetically engineered HyperAcute-Prostate cancer vaccine. It will establish the proper vaccine dose and will examine side effects and potential benefits of the treatment. The vaccine contains killed prostate cancer cells containing a mouse gene that causes the production of a foreign pattern of protein-sugars on the cell surface. It is hoped that the immune response to the foreign substance will stimulate the immune system to attack the patient's own cancer cells that have similar proteins without this sugar pattern, causing the tumor to remain stable or shrink.

Patients 19 years of age or older with hormone refractory prostate cancer that has recurred or no longer responds to standard treatment may be eligible for this study. Candidates will be screened with medical history and physical examination, blood tests, urinalysis, chest x-rays and CT scans. MRI, PET, and ultrasound scans may be obtained if needed.

Participants will receive twelve vaccinations two weeks apart from each other. The vaccines will be injected under the skin, similar to the way a tuberculosis skin test is given. Phase I of the study will treat successive groups of patients with increasing numbers of the vaccine cells to evaluate side effects of the treatment and determine the optimum dose. Phase II will look for any beneficial effects of the vaccine given at the highest dose found to be safe in Phase I. Monthly blood samples will be drawn during the 6 months of vaccine treatment. In addition, patient follow-up visits will be scheduled every 2 months for the remaining first year (6 months) after vaccination and then every 3 months for the next 2 years for the following tests and procedures to evaluate treatment response and side effects:

* Medical history and physical examination
* Blood tests
* X-rays and various scans (nuclear medicine/CT/MRI)
* FACT-P Assessment questionnaire to measure the impact of treatment on the patient's general well-being. The questionnaire is administered before beginning treatment, monthly during treatment, and during follow-up visits after completing the treatment. It includes questions on the severity of prostate cancer symptoms and the ability to perform normal activities of daily life.

DETAILED DESCRIPTION:
Prostate cancer is the most common type of cancer found in American men, other than skin cancer. The American Cancer Society estimated that there were about 230,900 new cases of prostate cancer in the United States in the year 2004. About 29,900 men will die of this disease. Prostate cancer is the second leading cause of cancer death in men, exceeded only by lung cancer. This protocol attempts to exploit an approach to prostate cancer immunotherapy using a naturally occurring barrier to xenotransplantation in humans in an attempt to vaccinate patients against their prostate cancer. The expression of the murine alpha (1,3) galactosyltransferase [alpha (1,3) GT] gene results in the cell surface expression of alpha (1,3) galactosyl-epitopes (alpha-gal) on membrane glycoproteins and glycolipids. These epitopes are the major target of the hyperacute rejection response that occurs when organs are transplanted from non-primate donor species into man. Human hosts often have pre-existing anti-alpha-gal antibodies that bind alpha-gal epitopes and lead to rapid activation of complement and cell lysis. The pre-existing anti-alpha-gal antibodies found in most individuals are thought to be due to exposure to alpha-gal epitopes that are naturally expressed on normal gut flora leading to chronic immunological stimulation. These antibodies may comprise up to 1% of serum IgG. In this Phase I/II trial, patients with hormone refractory prostate cancer will undergo a series of twelve intradermal injections with a vaccine composed of irradiated allogeneic prostate cancer cell lines (HAP-1 and HAP-2) that have been transduced with a recombinant Moloney murine leukemia virus (MoMLV)-based retroviral vector expressing the murine alpha (1,3) GT gene. Endpoints of the study include determination of dose-limiting toxicity (DLT), maximum tolerated dose (MTD), tumor and immunological responses.

ELIGIBILITY:
Inclusion Criteria:

* Phase I and Phase II Arm A: A histological diagnosis of prostate cancer with evidence of metastatic disease by CT scan or bone scan. Phase II, Arm B: Evidence of hormone refractive progressive disease by increasing PSA only.
* For patients enrolling in Phase II, Arm B: refractory to hormone therapy defined by: two consecutive increases in PSA documented over a previous reference value, the first occurring a minimum of 1 week from the reference value, with one value of at least 4 ng/mL and the increase(s) must be by at least 1.0 ng/mL.
* Castrate testosterone levels < 50 ng/dl (0.50 ng/mL)
* AJCC Stage IV (any T, any N, M1), hormone refractory metastatic, progressive or recurrent prostate carcinoma. Patients must have failed one attempt at hormonal therapy and may have received 2 prior chemotherapy regimens.
* ECOG performance status less than or equal to 2.
* Serum albumin greater than or equal to 3.0 gm/dL.
* Expected survival greater than or equal to 6 months.
* Subjects must have a negative serology for Hep B, C, and HIV prior to entering study.
* Adequate organ function including:

Marrow: *Hemoglobin greater than or equal to 10.0 mg/dL, *absolute granulocyte count (AGC) greater than or equal to 1,500/mm(3), *platelets greater than or equal to 100,000/mm(3), *absolute lymphocyte count greater than or equal to 475/mm(3).

Hepatic: *serum total bilirubin less than or equal to 1.5 x upper limit of normal (ULN), *ALT (SGPT) and AST (SGOT) less than or equal to 2.5 x ULN.

Renal: *serum creatinine less than or equal to 2.0 x ULN or creatinine clearance greater than or equal to 30 mL/min.

* All on-study tests must be less than or equal to Grade I toxicity for patient to be eligible for study, excluding serum LDH levels. PT, PTT must be less than or equal to 1.5 x ULN except for patients who are on therapeutic anticoagulant therapy.
* Measurable or bone metastases (Phase I, Phase II-Arm A) or non-measurable disease (Phase II-Arm B).
* Patients must have been treated with hormonal therapy and may have been treated with surgery and/or radiation therapy and/or less than or equal to 2 different chemotherapy regimens (including neoadjuvant and adjuvant treatment).
* Patients must be greater than or equal to 4 weeks since major surgery, radiotherapy, chemotherapy (6-weeks if they were treated with a nitrosourea or mitomycin) and recovered from the toxicity of prior treatment to less than or equal to Grade 1, exclusive of alopecia or fatigue.
* Patients must have the ability to understand the study, its risks, side effects, potential benefits and is able to give written informed consent to participate. Patients may not be consented by a durable power of attorney (DPA).
* Male subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental drug, and for one month after the last immunization.
* Patients taking bisphosphonates at the time of registration into the trial are eligible, but bisphosphonates must be continued at a constant level throughout the trial period. Bisphosphonate use must be initiated at least 28 days prior to first treatment.

Exclusion Criteria:

* Age less than 19 years of age.
* Active CNS metastases or carcinomatous meningitis.
* Hypercalcemia greater than 2.9 mmol/L, unresponsive to standard therapy.
* Other malignancy within last 5 years, unless the probability of recurrence of the prior malignancy is less than 5%. Patients curatively treated for squamous and basal cell carcinoma of the skin or patients with a history of malignant tumor in the past that have been disease free for at least 5 years are also eligible for this study.
* History of organ transplant or active immunosuppressive therapy (such as cyclosporine, tacrolimus, etc.).
* Subjects taking systemic corticosteroid therapy for any reason are not eligible.
* Significant or uncontrolled congestive heart failure, myocardial infarction or significant ventricular arrhythmias within the last six months.
* Active infection or antibiotics within 1-week prior to study, including unexplained fever (temp. greater than 38.1 degrees Celsius).
* Autoimmune disease (e.g., systemic lupus erythematosis, active rheumatoid arthritis, etc). Patients with a remote history of asthma or mild active asthma are eligible.
* Other serious medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis).
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc).
* A known allergy to any component of the alpha (1,3) galactosyltransferase tumor vaccine or cell lines from which it is derived.
* Concurrent therapy such as palliative radiation or opioid analgesics for tumor-associated pain.
* Anti-androgen therapy within 42 days of first treatment.
* Treatment with cimetidine within 30 days of first treatment.
* Prior splenectomy.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of administration of HyperAcute-Prostate (HAP) cancer cells by injection into men with hormone refractory prostate carcinoma | 6 months

SECONDARY OUTCOMES:
Correlative scientific studies of patient samples to determine the mechanism of any observed anti-tumor effect | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles J. Link, M.D., Study Chair — NewLink Genetics Corporation
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States